CLINICAL TRIAL: NCT04572893
Title: An Open-Label, Exploratory Study of the Safety and Preliminary Efficacy of Danicamtiv in Stable Ambulatory Participants With Primary Dilated Cardiomyopathy Due to Either MYH7 or TTN Variants or Other Causalities
Brief Title: Exploratory Study of Danicamtiv in Patients With Primary Dilated Cardiomyopathy (DCM) Due to Genetic Variants or Other Causalities
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CV028-005; 2019-003626-24 (EudraCT Number)
Record Dates: First submitted 2020-09-09; First posted 2020-10-01 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Primary Familial Dilated Cardiomyopathy
Keywords: Primary dilated cardiomyopathy (DCM); Familial dilated cardiomyopathy (DCM); Myosin Heavy Chain 7 (MYH7); Titin (TTN); MYK-491; danicamtiv
MeSH Terms: conditions — Campomelic Dysplasia; Cardiomyopathy, Dilated; familial dilated cardiomyopathy; Distal Myopathies; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MYK-491 (Experimental): Primary DCM due to MYH7 or TTN Variant or due to other causalities not related to MYH7 or TTN variants
  Interventions: Drug: danicamtiv

INTERVENTIONS:
Drug: danicamtiv — Myosin activator
  Other Names: MYK-491; BMS-986434

SUMMARY:
The purpose of this Phase 2a study is to establish safety and preliminary efficacy of treatment with danicamtiv in patients with primary dilated cardiomyopathy (DCM) due to MYH7 or TTN variants or other causalities.

ELIGIBILITY:
Inclusion Criteria:

* For MYH7 and TTN cohorts, must have diagnosis of primary DCM (dilated cardiomyopathy), clinically stable and due to probably disease-causing variant of MYH7 or TTN
* Has adequate acoustic windows for echocardiography
* Maximum of 3 family members with same variant can be enrolled
* For the cohort of primary DCM due to causalities other than MYH7 and TTN, participant must have diagnosis of primary DCM with a cause not related to MYH7 or TTN variants

Exclusion Criteria:

* Significant structural cardiac abnormalities including valvar dysfunction on Screening transthoracic echo(s)
* Routinely scheduled outpatient intravenous (IV) infusions for heart failure (e.g., inotropes, afterload reduction, or diuretics)
* Presence of protocol specified laboratory abnormalities at Screening
* Recent acute coronary syndrome or angina pectoris (<90 days)
* Recent hospitalization for heart failure (<90 days)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (19):
- United States (12):
  - Local Institution - 0007, La Jolla, California
  - Local Institution - 0010, Washington D.C., District of Columbia
  - Local Institution - 0009, Tampa, Florida
  - Local Institution - 0002, Chicago, Illinois
  - Local Institution - 0003, Boston, Massachusetts
  - Local Institution - 0005, Rochester, Minnesota
  - Local Institution - 0006, Cleveland, Ohio
  - Local Institution - 0019, Columbus, Ohio
  - Local Institution - 0001, Philadelphia, Pennsylvania
  - Local Institution - 0004, Charleston, South Carolina
  - Local Institution - 0008, Germantown, Tennessee
  - Local Institution - 0018, Austin, Texas
- Germany (2):
  - Local Institution - 0014, Heidelberg, Baden-Wurttemberg
  - Local Institution - 0015, Würzburg
- Spain (3):
  - Local Institution - 0012, A Coruña
  - Local Institution - 0011, El Palmar
  - Local Institution - 0013, Majadahonda
- United Kingdom (2):
  - Local Institution - 0016, London
  - Local Institution - 0017, Middlesex

REFERENCES:
- [Derived] Lakdawala NK, Hershberger RE, Garcia-Pavia P, Elliott PM, Ginns J, Meder B, Solomon S, Cunningham JW, Gimeno JR, Barriales-Villa R, Adler E, Gerull B, Pereira NL, Halliday BP, Li W, Jarugula P, Maruyama S, Mohran SE, Papadaki M, Anto AR, Anderson RL, Rodriguez HM, Del Rio CL, Edelberg JM, Kurio G, Maya J, Januzzi JL. Danicamtiv, a Selective Agonist of Cardiac Myosin, for Dilated Cardiomyopathy: A Phase 2 Open-Label Trial. J Am Coll Cardiol. 2025 Dec 23;86(25):2598-2612. doi: 10.1016/j.jacc.2025.09.1511. Epub 2025 Sep 29. PMID 41217321
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part B will commence after a participant completes Part A and opts to continue onto Part B. Individual participant doses for Part B will be based on systolic ejection time increase in Part A.
Groups:
- Part A - MYH7 - MYK-491: Participants with myosin heavy chain 7 (MYH7) variant received Danicamtiv. Study drug will be administered orally BID for at least 5 days and up to 8 days for each Treatment Period
- Part A - TTN - MYK-491: Participants with titin (TTN) variant received Danicamtiv. Study drug will be administered orally BID for at least 5 days and up to 8 days for each Treatment Period
- Part A - DCM-Genetic - MYK-491: Participants with dilated cardiomyopathy (DCM)-Genetic received Danicamtiv. Study drug will be administered orally BID for at least 5 days and up to 8 days for each Treatment Period
- Part A - DCM-Non Genetic - MYK-491: Participants with dilated cardiomyopathy (DCM)-Non genetic received Danicamtiv. Study drug will be administered orally BID for at least 5 days and up to 8 days for each Treatment Period
- Part B - MYH7 - MYK-491: Participants with MYH7 variant received Danicamtiv after meeting eligibility criteria
- Part B - TTN - MYK-491: Participants with TTN variant received Danicamtiv after meeting eligibility criteria
- Part B - DCM-Non Genetic - MYK-491: Participants with DCM-Non genetic received Danicamtiv after meeting eligibility criteria
Period: Part A
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491 | Part B - MYH7 - MYK-491 | Part B - TTN - MYK-491 | Part B - DCM-Non Genetic - MYK-491
Started | 12 | 14 | 5 | 10 | 0 | 0 | 0
Started Part B | 8 | 7 | 0 | 4 | 0 | 0 | 0
Completed | 11 | 14 | 5 | 10 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491 | Part B - MYH7 - MYK-491 | Part B - TTN - MYK-491 | Part B - DCM-Non Genetic - MYK-491
Started | 0 | 0 | 0 | 0 | 8 | 7 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 8 | 7 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 7 | 5 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491 | Total
Number analyzed (Participants) | 12 | 14 | 5 | 10 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 4 | 9 | 36
  >=65 years | 1 | 2 | 1 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 2 | 2 | 15
  Male | 5 | 10 | 3 | 8 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 1 | 0 | 5
  Not Hispanic or Latino | 9 | 13 | 3 | 10 | 35
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 0 | 0 | 0 | 1
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 2
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 11 | 14 | 5 | 8 | 38
  Uknown | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) in Part A
Description: An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first dose to 30 days post last dose (Up to approximately 15 weeks)
Population: All treated participants in Part A as pre-specified in protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 12 | 14 | 5 | 10
Participants | 9 | 9 | 4 | 4

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) in Part A
Description: An SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability or permanent damage, is a congenital anomaly/birth defect, is an important medical event.
Time Frame: From first dose to 30 days post last dose (Up to approximately 15 weeks)
Population: All treated participants in Part A as pre-specified in protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 12 | 14 | 5 | 10
Participants | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Safety Laboratory Assessments by Intensity in Part A
Description: Number of participants with safety laboratory assessments by intensity. Mild=An event that is easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities; Moderate= An event causing sufficient discomfort and interferes with normal everyday activities.
Time Frame: From first dose to 14 days post last dose (Up to approximately 13 weeks)
Population: All treated participants in Part A as pre-specified in protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 12 | 14 | 5 | 10
Participants
  Alanine aminotransferase increased Mild | 1 | 0 | 1 | 0
  Aspartate aminotransferase increased Mild | 1 | 0 | 1 | 0
  Blood creatinine increased Moderate | 0 | 0 | 1 | 0
  Fibrin D dimer increased Moderate | 0 | 1 | 0 | 0
  Hyperkalaemia Mild | 0 | 1 | 0 | 0
  Hyperkalaemia Moderate | 0 | 0 | 1 | 0

4. Secondary Outcome: Transthoracic Echo (TTE) Left Ventricular Ejection Time (LVET) Change From Baseline
Description: Baseline is defined as the last non-missing result prior to the first dose of study medication. for part B, baseline is defined as visit 1B regardless of rescreening. Treatment periods 1 and 2 are 5 to 8 days.
Time Frame: Part A: Baseline, end of treatment period 1. end of treatment period 2, early termination; Part B: Baseline, weeks 2, 6, 12, 24, 36, 48, and early termination
Population: All treated participants with baseline and post baseline measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: msec
Groups:
- Part B - MYH7 - MYK-491: Participants with MYH7 variant received Danicamtiv orally BID after meeting eligibility criteria
- Part B - TTN - MYK-491: Participants with TTN variant received Danicamtiv orally BID after meeting eligibility criteria
- Part B - DCM-Non Genetic - MYK-491: Participants with DCM-Non genetic received Danicamtiv orally BID after meeting eligibility criteria
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491 | Part B - MYH7 - MYK-491 | Part B - TTN - MYK-491 | Part B - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 12 | 14 | 5 | 10 | 8 | 7 | 4
msec
  End of treatment period 1: number analyzed (Participants) | 12 | 14 | 4 | 10 | 0 | 0 | 0
  End of treatment period 1 | 12.1 (23.7) | 7.4 (28.8) | -3.5 (8.7) | 3.3 (36.3) |  |  |
  End of treatment period 2: number analyzed (Participants) | 11 | 14 | 5 | 10 | 0 | 0 | 0
  End of treatment period 2 | 29.4 (31.0) | 29.0 (25.4) | -5.6 (18.2) | 15.2 (54.4) |  |  |
  week 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 7 | 4
  week 2 |  |  |  |  | 38.3 (30.0) | 44.3 (16.3) | 20.3 (34.5)
  week 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 6 | 2
  week 6 |  |  |  |  | 25.3 (22.3) | 53.3 (43.6) | 20.5 (67.2)
  week 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 6 | 1
  week 12 |  |  |  |  | 32.1 (27.4) | 38.2 (33.5) | 44.0 (NA) — Insufficient number of participants to calculate standard deviation
  week 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 5 | 0
  week 24 |  |  |  |  | 39.8 (46.3) | 59.8 (39.5) |
  week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 2 | 0
  week 36 |  |  |  |  |  | 47.5 (9.2) |
  week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 4 | 0
  week 48 |  |  |  |  | 42.3 (40.3) | 30.3 (34.0) |
  Early termination: number analyzed (Participants) | 1 | 0 | 0 | 0 | 8 | 7 | 3
  Early termination | -23.0 (NA) — Insufficient number of participants to calculate standard deviation |  |  |  | 13.5 (44.4) | -1.4 (20.5) | -14.3 (35.2)

5. Primary Outcome: Number of Participants With Clinically Significant Changes in Physical Examinations in Part A
Description: Number of participants with clinically significant changes in physical examinations.
Time Frame: From first dose to 30 days post last dose (Up to approximately 15 weeks)
Population: All treated participants in Part A as pre-specified in protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 12 | 14 | 5 | 10
Participants | 0 | 1 | 0 | 0

6. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs in Part A
Description: Number of participants with clinically significant changes in vital signs.
Time Frame: From first dose to 30 days post last dose (Up to approximately 15 weeks)
Population: All treated participants in Part A as pre-specified in protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 12 | 14 | 5 | 10
Participants | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Clinically Significant Changes in 12-Lead ECG Recordings in Part A
Description: Number of participants with clinically significant changes in 12-lead ECG recordings.
Time Frame: From first dose to 30 days post last dose (Up to approximately 15 weeks)
Population: All treated participants in Part A as pre-specified in protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 12 | 14 | 5 | 10
Participants | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) by Intensity in Part A
Description: An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment.
  Mild=An event that is easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities; Moderate= An event causing sufficient discomfort and interferes with normal everyday activities.
  Severe= An event preventing normal everyday activities. (An AE that is assessed as severe should not be confused with a SAE. Severe is a category utilized for rating the intensity of an event; and both AEs and SAEs can be assessed as severe.)
Time Frame: From first dose to 14 days post last dose (Up to approximately 13 weeks)
Population: All treated participants in Part A as pre-specified in protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 12 | 14 | 5 | 10
Participants
  Mild | 8 | 6 | 3 | 4
  Moderate | 0 | 1 | 1 | 0
  Severe | 0 | 0 | 0 | 0

9. Secondary Outcome: Transthoracic Echo (TTE) Left Ventricular Stroke Volume (LVSV) Change From Baseline
Description: as for outcome 4
Time Frame: as for outcome 4
Population: All treated participants with baseline and post baseline measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491 | Part B - MYH7 - MYK-491 | Part B - TTN - MYK-491 | Part B - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 11 | 14 | 5 | 10 | 8 | 7 | 4
mL
  End of treatment period 1: number analyzed (Participants) | 11 | 13 | 4 | 9 | 0 | 0 | 0
  End of treatment period 1 | 10.581 (9.814) | 5.628 (3.127) | 1.855 (7.979) | -5.897 (17.237) |  |  |
  End of treatment period 2: number analyzed (Participants) | 11 | 14 | 5 | 10 | 0 | 0 | 0
  End of treatment period 2 | 10.151 (19.585) | 1.243 (14.275) | 1.050 (13.379) | 2.172 (20.000) |  |  |
  week 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 7 | 4
  week 2 |  |  |  |  | 15.576 (11.932) | -7.600 (14.358) | -15.678 (18.882)
  week 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 6 | 1
  week 6 |  |  |  |  | 7.778 (21.508) | 18.313 (14.697) | 16.500 (NA) — Insufficient number of participants to calculate standard deviation
  week 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 4 | 1
  week 12 |  |  |  |  | 19.410 (21.832) | 24.853 (18.181) | 22.320 (NA) — Insufficient number of participants to calculate standard deviation
  week 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 5 | 0
  week 24 |  |  |  |  | 13.893 (14.892) | 25.174 (24.052) |
  week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  week 36 |  |  |  |  |  | -20.450 (NA) — Insufficient number of participants to calculate standard deviation |
  week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 3 | 0
  week 48 |  |  |  |  | 19.070 (16.317) | -6.863 (12.464) |
  Early termination: number analyzed (Participants) | 1 | 0 | 0 | 0 | 8 | 7 | 3
  Early termination | 0.650 (NA) — Insufficient number of participants to calculate standard deviation |  |  |  | 2.684 (30.133) | -11.136 (14.539) | 5.533 (20.941)

10. Secondary Outcome: Transthoracic Echo (TTE) Left Ventricular Ejection Fraction (LVEF) Change From Baseline
Description: as for outcome 4
Time Frame: Part A: Baseline, end of treatment period 1. end of treatment period 2, early termination; Part B: Baseline, weeks 2, 6, 12, 24, 36, 42, 48, and early termination
Population: All treated participants with baseline and post baseline measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491 | Part B - MYH7 - MYK-491 | Part B - TTN - MYK-491 | Part B - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 12 | 14 | 4 | 10 | 8 | 7 | 3
percentage
  End of treatment period 1: number analyzed (Participants) | 12 | 14 | 4 | 10 | 0 | 0 | 0
  End of treatment period 1 | 4.78 (7.40) | 4.94 (7.08) | -0.75 (3.06) | 2.47 (6.14) |  |  |
  End of treatment period 2: number analyzed (Participants) | 11 | 13 | 4 | 9 | 0 | 0 | 0
  End of treatment period 2 | 8.84 (6.43) | 5.94 (6.15) | 1.37 (5.36) | 4.84 (10.00) |  |  |
  week 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 7 | 2
  week 2 |  |  |  |  | 5.53 (10.31) | 4.21 (11.03) | 5.60 (2.12)
  week 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 6 | 2
  week 6 |  |  |  |  | 3.31 (5.85) | -0.40 (7.83) | 14.05 (18.03)
  week 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 6 | 1
  week 12 |  |  |  |  | 2.44 (5.39) | 1.77 (5.26) | 7.60 (NA) — Insufficient number of participants to calculate standard deviation
  week 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 5 | 0
  week 24 |  |  |  |  | -2.78 (0.59) | 2.24 (8.58) |
  week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  week 36 |  |  |  |  |  | 10.80 (NA) — Insufficient number of participants to calculate standard deviation |
  Week 42: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Week 42 |  |  |  |  |  | 23.60 (NA) — Insufficient number of participants to calculate standard deviation |
  week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 4 | 0
  week 48 |  |  |  |  | 3.85 (4.75) | 7.12 (11.12) |
  Early termination: number analyzed (Participants) | 1 | 0 | 0 | 0 | 8 | 7 | 3
  Early termination | -3.20 (NA) — Insufficient number of participants to calculate standard deviation |  |  |  | -2.94 (4.65) | 3.99 (9.55) | 4.13 (5.87)

11. Secondary Outcome: Transthoracic Echo (TTE) Left Ventricular Global Longitudinal Strain (LVGLS) Change From Baseline
Description: as for outcome 4
Time Frame: as for outcome 10
Population: All treated participants with baseline and post baseline measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491 | Part B - MYH7 - MYK-491 | Part B - TTN - MYK-491 | Part B - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 12 | 14 | 5 | 10 | 8 | 7 | 4
percentage
  End of treatment period 1: number analyzed (Participants) | 12 | 14 | 4 | 10 | 0 | 0 | 0
  End of treatment period 1 | -1.41 (2.79) | -0.79 (2.31) | -0.32 (2.81) | -0.36 (1.63) |  |  |
  End of treatment period 2: number analyzed (Participants) | 11 | 14 | 5 | 10 | 0 | 0 | 0
  End of treatment period 2 | -2.05 (2.05) | -1.21 (2.23) | -1.92 (2.00) | -0.95 (2.46) |  |  |
  week 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 7 | 4
  week 2 |  |  |  |  | -1.60 (2.59) | -1.84 (1.66) | -1.80 (2.63)
  week 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 6 | 2
  week 6 |  |  |  |  | -2.18 (2.53) | -1.90 (1.11) | -3.65 (0.49)
  week 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 6 | 1
  week 12 |  |  |  |  | -2.34 (2.03) | -2.00 (2.34) | -4.00 (NA) — Insufficient number of participants to calculate standard deviation
  week 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 5 | 0
  week 24 |  |  |  |  | 0.02 (1.25) | -2.62 (2.66) |
  week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  week 36 |  |  |  |  |  | -2.50 (NA) — Insufficient number of participants to calculate standard deviation |
  Week 42: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Week 42 |  |  |  |  |  | -7.70 (NA) — Insufficient number of participants to calculate standard deviation |
  week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 4 | 0
  week 48 |  |  |  |  | -2.77 (1.99) | -4.33 (1.30) |
  Early termination: number analyzed (Participants) | 1 | 0 | 0 | 0 | 8 | 7 | 3
  Early termination | -0.70 (NA) — Insufficient number of participants to calculate standard deviation |  |  |  | 0.01 (2.12) | -1.31 (1.41) | -1.90 (1.81)

12. Secondary Outcome: Transthoracic Echo (TTE) Left Ventricular Global Circumferential Strain (LVGCS) Change From Baseline
Description: as for outcome 4
Time Frame: as for outcome 10
Population: All treated participants with baseline and post baseline measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491 | Part B - MYH7 - MYK-491 | Part B - TTN - MYK-491 | Part B - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 10 | 10 | 4 | 10 | 7 | 7 | 4
percentage
  End of treatment period 1: number analyzed (Participants) | 10 | 10 | 3 | 10 | 0 | 0 | 0
  End of treatment period 1 | -3.62 (3.73) | 0.58 (2.83) | -4.10 (4.07) | 0.15 (4.47) |  |  |
  End of treatment period 2: number analyzed (Participants) | 10 | 10 | 4 | 10 | 0 | 0 | 0
  End of treatment period 2 | -4.00 (3.17) | -1.45 (3.32) | -2.08 (1.25) | -0.78 (3.87) |  |  |
  week 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 7 | 4
  week 2 |  |  |  |  | -5.16 (4.55) | -3.00 (3.64) | -3.25 (5.30)
  week 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 5 | 1
  week 6 |  |  |  |  | -4.07 (3.43) | -4.68 (1.11) | -0.10 (NA) — Insufficient number of participants to calculate standard deviation
  week 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 5 | 1
  week 12 |  |  |  |  | -3.80 (1.26) | -0.94 (2.65) | 0.00 (NA) — Insufficient number of participants to calculate standard deviation
  week 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 5 | 0
  week 24 |  |  |  |  | -2.64 (4.72) | -0.88 (1.94) |
  week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  week 36 |  |  |  |  |  | -2.60 (NA) — Insufficient number of participants to calculate standard deviation |
  Week 42: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Week 42 |  |  |  |  |  | -6.00 (NA) — Insufficient number of participants to calculate standard deviation |
  week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 4 | 0
  week 48 |  |  |  |  | -4.05 (3.13) | -3.98 (3.43) |
  Early termination: number analyzed (Participants) | 1 | 0 | 0 | 0 | 7 | 6 | 2
  Early termination | 0.40 (NA) — Insufficient number of participants to calculate standard deviation |  |  |  | 0.54 (5.50) | -1.52 (2.38) | 0.40 (5.23)

13. Secondary Outcome: Transthoracic Echo (TTE) Tissue Doppler Imaging (TDI) S Prime Lateral Change From Baseline
Description: as for outcome 4
Time Frame: as for outcome 4
Population: All treated participants with baseline and post baseline measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491 | Part B - MYH7 - MYK-491 | Part B - TTN - MYK-491 | Part B - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 11 | 13 | 5 | 10 | 8 | 7 | 2
cm/s
  End of treatment period 1: number analyzed (Participants) | 11 | 13 | 4 | 9 | 0 | 0 | 0
  End of treatment period 1 | 0.23 (1.90) | -0.12 (0.77) | 1.15 (0.66) | 0.22 (1.62) |  |  |
  End of treatment period 2: number analyzed (Participants) | 11 | 12 | 5 | 10 | 0 | 0 | 0
  End of treatment period 2 | 1.01 (1.75) | 0.53 (1.57) | 1.40 (1.38) | -0.10 (1.99) |  |  |
  week 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 7 | 2
  week 2 |  |  |  |  | -0.04 (1.62) | -0.14 (0.88) | -0.95 (0.78)
  week 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 6 | 1
  week 6 |  |  |  |  | 0.34 (0.84) | 0.08 (0.59) | -0.80 (NA) — Insufficient number of participants to calculate standard deviation
  week 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 6 | 0
  week 12 |  |  |  |  | 0.57 (1.26) | -0.03 (1.29) |
  week 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 5 | 0
  week 24 |  |  |  |  | -0.55 (1.33) | 0.18 (0.65) |
  week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  week 36 |  |  |  |  |  | -0.30 (NA) — Insufficient number of participants to calculate standard deviation |
  week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 3 | 0
  week 48 |  |  |  |  | 1.25 (1.35) | 0.10 (0.46) |
  Early termination: number analyzed (Participants) | 1 | 0 | 0 | 0 | 8 | 7 | 2
  Early termination | -2.30 (NA) — Insufficient number of participants to calculate standard deviation |  |  |  | 0.14 (1.43) | 0.67 (1.39) | -1.20 (0.57)

14. Secondary Outcome: Transthoracic Echo (TTE) Tissue Doppler Imaging (TDI) S Prime Septal Change From Baseline
Description: as for outcome 4
Time Frame: as for outcome 4
Population: All treated participants with baseline and post baseline measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491 | Part B - MYH7 - MYK-491 | Part B - TTN - MYK-491 | Part B - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 12 | 13 | 5 | 10 | 8 | 7 | 3
cm/s
  End of treatment period 1: number analyzed (Participants) | 12 | 12 | 4 | 9 | 0 | 0 | 0
  End of treatment period 1 | 0.56 (1.05) | 0.03 (0.50) | 0.78 (0.63) | 0.06 (0.66) |  |  |
  End of treatment period 2: number analyzed (Participants) | 11 | 13 | 5 | 10 | 0 | 0 | 0
  End of treatment period 2 | 0.53 (0.42) | 0.20 (0.62) | 1.04 (1.57) | -0.20 (0.94) |  |  |
  week 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 7 | 3
  week 2 |  |  |  |  | 0.24 (0.90) | 0.06 (0.58) | 0.20 (1.31)
  week 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 6 | 2
  week 6 |  |  |  |  | 0.95 (0.89) | 0.50 (1.39) | -0.05 (1.34)
  week 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 6 | 1
  week 12 |  |  |  |  | 0.77 (0.83) | -0.12 (0.74) | 1.30 (NA) — Insufficient number of participants to calculate standard deviation
  week 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 4 | 0
  week 24 |  |  |  |  | 0.17 (0.53) | 0.17 (0.97) |
  week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  week 36 |  |  |  |  |  | -1.40 (NA) — Insufficient number of participants to calculate standard deviation |
  week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 3 | 0
  week 48 |  |  |  |  | 1.22 (1.27) | 0.07 (1.14) |
  Early termination: number analyzed (Participants) | 1 | 0 | 0 | 0 | 8 | 7 | 3
  Early termination | 0.40 (NA) — Insufficient number of participants to calculate standard deviation |  |  |  | 0.40 (1.53) | 0.10 (0.77) | 0.67 (1.00)

15. Secondary Outcome: Transthoracic Echo (TTE) Tissue Doppler Imaging (TDI) Left Ventricular End-Systolic Diameter (LVESD) Change From Baseline
Description: as for outcome 4
Time Frame: as for outcome 4
Population: All treated participants with baseline and post baseline measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491 | Part B - MYH7 - MYK-491 | Part B - TTN - MYK-491 | Part B - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 12 | 13 | 5 | 10 | 7 | 7 | 3
mm
  End of treatment period 1: number analyzed (Participants) | 12 | 13 | 5 | 7 | 0 | 0 | 0
  End of treatment period 1 | -0.15 (4.07) | -2.84 (3.47) | 0.10 (1.44) | -1.77 (5.60) |  |  |
  End of treatment period 2: number analyzed (Participants) | 11 | 13 | 5 | 10 | 0 | 0 | 0
  End of treatment period 2 | -3.14 (5.97) | -5.48 (4.83) | -3.60 (3.48) | -2.20 (6.03) |  |  |
  week 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 7 | 3
  week 2 |  |  |  |  | -0.90 (4.25) | -5.94 (3.74) | -4.43 (9.40)
  week 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 6 | 1
  week 6 |  |  |  |  | -0.17 (6.01) | -5.93 (4.76) | -2.20 (NA) — Insufficient number of participants to calculate standard deviation
  week 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 6 | 1
  week 12 |  |  |  |  | -0.92 (4.67) | -4.18 (4.75) | -1.60 (NA) — Insufficient number of participants to calculate standard deviation
  week 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 5 | 0
  week 24 |  |  |  |  | -0.07 (6.04) | -6.12 (4.18) |
  week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  week 36 |  |  |  |  |  | -5.80 (NA) — Insufficient number of participants to calculate standard deviation |
  week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 4 | 0
  week 48 |  |  |  |  | 2.90 (7.07) | -4.90 (3.53) |
  Early termination: number analyzed (Participants) | 1 | 0 | 0 | 0 | 7 | 7 | 3
  Early termination | -1.50 (NA) — Insufficient number of participants to calculate standard deviation |  |  |  | 1.33 (10.57) | -0.77 (3.86) | -0.60 (5.36)

16. Secondary Outcome: Transthoracic Echo (TTE) Tissue Doppler Imaging (TDI) Left Ventricular End-Systolic Volumen Index (LVESVi) Change From Baseline
Description: as for outcome 4
Time Frame: as for outcome 10
Population: All treated participants with baseline and post baseline measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491 | Part B - MYH7 - MYK-491 | Part B - TTN - MYK-491 | Part B - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 12 | 14 | 4 | 10 | 8 | 7 | 3
mL/m^2
  End of treatment period 1: number analyzed (Participants) | 12 | 14 | 4 | 10 | 0 | 0 | 0
  End of treatment period 1 | -8.3128 (9.2045) | -2.8341 (10.6672) | 1.5998 (2.6613) | -3.1748 (6.3863) |  |  |
  End of treatment period 2: number analyzed (Participants) | 11 | 13 | 4 | 9 | 0 | 0 | 0
  End of treatment period 2 | -9.0315 (10.6354) | -7.0016 (8.8423) | -1.7459 (6.9756) | -4.3387 (8.9773) |  |  |
  week 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 7 | 2
  week 2 |  |  |  |  | -16.6661 (27.1117) | -6.1675 (12.9178) | -3.7087 (2.2142)
  week 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 6 | 2
  week 6 |  |  |  |  | -6.8323 (14.6055) | -7.9134 (10.2267) | -13.2403 (18.8755)
  week 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 6 | 1
  week 12 |  |  |  |  | -5.5205 (9.5934) | -9.9285 (14.1805) | -0.9776 (NA) — Insufficient number of participants to calculate standard deviation
  week 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 5 | 0
  week 24 |  |  |  |  | -2.2674 (14.6852) | -6.6309 (19.3049) |
  week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 2 | 0
  week 36 |  |  |  |  |  | -21.4681 (6.5099) |
  Week 42: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Week 42 |  |  |  |  |  | -29.9173 (NA) — Insufficient number of participants to calculate standard deviation |
  week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 4 | 0
  week 48 |  |  |  |  | -13.5827 (21.5043) | -18.4947 (12.9649) |
  Early termination: number analyzed (Participants) | 1 | 0 | 0 | 0 | 8 | 7 | 3
  Early termination | 1.2208 (NA) — Insufficient number of participants to calculate standard deviation |  |  |  | -2.3523 (14.4189) | -6.7128 (15.2440) | 2.9170 (6.0452)

17. Secondary Outcome: Transthoracic Echo (TTE) Tissue Doppler Imaging (TDI) Left Ventricular End-Diastolic Diameter (LVEDD) Change From Baseline
Description: as for outcome 4
Time Frame: as for outcome 4
Population: All treated participants with baseline and post baseline measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491 | Part B - MYH7 - MYK-491 | Part B - TTN - MYK-491 | Part B - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 12 | 13 | 5 | 10 | 8 | 7 | 4
mm
  End of treatment period 1: number analyzed (Participants) | 12 | 13 | 5 | 9 | 0 | 0 | 0
  End of treatment period 1 | 0.48 (3.61) | -2.49 (3.51) | -0.60 (3.91) | -1.37 (5.14) |  |  |
  End of treatment period 2: number analyzed (Participants) | 11 | 13 | 5 | 10 | 0 | 0 | 0
  End of treatment period 2 | -0.85 (4.36) | -3.12 (3.34) | -3.50 (3.84) | -1.77 (4.60) |  |  |
  week 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 7 | 4
  week 2 |  |  |  |  | -5.11 (9.22) | -3.56 (4.03) | -5.00 (7.04)
  week 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 6 | 1
  week 6 |  |  |  |  | -1.75 (3.34) | -3.10 (2.61) | 0.30 (NA) — Insufficient number of participants to calculate standard deviation
  week 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 6 | 1
  week 12 |  |  |  |  | -2.09 (3.58) | -0.17 (2.64) | 0.90 (NA) — Insufficient number of participants to calculate standard deviation
  week 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 5 | 0
  week 24 |  |  |  |  | -2.10 (2.50) | -2.86 (5.87) |
  week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  week 36 |  |  |  |  |  | -3.10 (NA) — Insufficient number of participants to calculate standard deviation |
  Week 42: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Week 42 |  |  |  |  |  | -1.50 (NA) — Insufficient number of participants to calculate standard deviation |
  week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 4 | 0
  week 48 |  |  |  |  | -3.40 (3.64) | -2.13 (3.40) |
  Early termination: number analyzed (Participants) | 1 | 0 | 0 | 0 | 8 | 7 | 2
  Early termination | 3.60 (NA) — Insufficient number of participants to calculate standard deviation |  |  |  | -1.97 (5.36) | 0.46 (3.40) | 2.70 (1.13)

18. Secondary Outcome: Transthoracic Echo (TTE) Tissue Doppler Imaging (TDI) Left Ventricular End-Diastolic Volumen Index (LVEDVi) Change From Baseline
Description: as for outcome 4
Time Frame: as for outcome 10
Population: All treated participants with baseline and post baseline measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: m1/m2
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491 | Part B - MYH7 - MYK-491 | Part B - TTN - MYK-491 | Part B - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 12 | 14 | 4 | 10 | 8 | 7 | 3
m1/m2
  End of treatment period 1: number analyzed (Participants) | 12 | 14 | 4 | 10 | 0 | 0 | 0
  End of treatment period 1 | -7.3006 (7.0043) | 0.4855 (10.8288) | 1.3937 (3.9810) | -3.6715 (8.4975) |  |  |
  End of treatment period 2: number analyzed (Participants) | 11 | 13 | 4 | 9 | 0 | 0 | 0
  End of treatment period 2 | -4.3719 (11.6238) | -4.4642 (12.9621) | -1.1050 (6.1575) | -2.1417 (12.8270) |  |  |
  week 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 7 | 2
  week 2 |  |  |  |  | -19.7184 (31.0876) | -6.7773 (10.3963) | 0.2596 (0.0152)
  week 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 6 | 2
  week 6 |  |  |  |  | -6.2694 (17.5060) | -12.9208 (11.0202) | -11.4771 (18.4933)
  week 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 6 | 1
  week 12 |  |  |  |  | -5.2247 (11.4301) | -11.7627 (17.1607) | 7.4828 (NA) — Insufficient number of participants to calculate standard deviation
  week 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 5 | 0
  week 24 |  |  |  |  | -5.9020 (20.7779) | -6.2700 (24.3104) |
  week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 2 | 0
  week 36 |  |  |  |  |  | -13.0453 (5.3813) |
  Week 42: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Week 42 |  |  |  |  |  | -11.8121 (NA) — Insufficient number of participants to calculate standard deviation |
  week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 4 | 0
  week 48 |  |  |  |  | -14.3351 (24.7973) | -18.5657 (6.0845) |
  Early termination: number analyzed (Participants) | 1 | 0 | 0 | 0 | 8 | 7 | 3
  Early termination | -1.6197 (NA) — Insufficient number of participants to calculate standard deviation |  |  |  | -7.2323 (24.2148) | -6.7050 (17.2581) | 8.3887 (3.3592)

19. Secondary Outcome: Transthoracic Echo (TTE) Tissue Doppler Imaging (TDI) E Prime Lateral Change From Baseline
Description: as for outcome 4
Time Frame: as for outcome 4
Population: All treated participants with baseline and post baseline measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491 | Part B - MYH7 - MYK-491 | Part B - TTN - MYK-491 | Part B - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 11 | 12 | 5 | 10 | 8 | 6 | 3
cm/s
  End of treatment period 1: number analyzed (Participants) | 11 | 12 | 4 | 8 | 0 | 0 | 0
  End of treatment period 1 | 0.55 (1.63) | 0.37 (2.51) | 1.23 (1.21) | 0.46 (3.27) |  |  |
  End of treatment period 2: number analyzed (Participants) | 11 | 11 | 5 | 10 | 0 | 0 | 0
  End of treatment period 2 | 0.51 (1.50) | 0.58 (2.97) | 2.60 (3.38) | -0.66 (2.23) |  |  |
  week 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 6 | 3
  week 2 |  |  |  |  | 0.23 (2.77) | 0.42 (1.47) | -1.30 (1.51)
  week 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 5 | 2
  week 6 |  |  |  |  | 0.43 (1.18) | -0.14 (1.29) | -1.30 (0.99)
  week 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 5 | 1
  week 12 |  |  |  |  | 0.83 (1.99) | -1.48 (2.36) | -3.20 (NA) — Insufficient number of participants to calculate standard deviation
  week 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 4 | 0
  week 24 |  |  |  |  | 0.15 (1.52) | -0.40 (2.09) |
  week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  week 36 |  |  |  |  |  | -1.80 (NA) — Insufficient number of participants to calculate standard deviation |
  week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 3 | 0
  week 48 |  |  |  |  | 2.25 (1.89) | -0.30 (1.60) |
  Early termination: number analyzed (Participants) | 1 | 0 | 0 | 0 | 8 | 6 | 3
  Early termination | -0.60 (NA) — Insufficient number of participants to calculate standard deviation |  |  |  | 0.20 (2.85) | 0.37 (2.28) | 2.23 (2.16)

20. Secondary Outcome: Transthoracic Echo (TTE) Tissue Doppler Imaging (TDI) E Prime Septal Change From Baseline
Description: as for outcome 4
Time Frame: as for outcome 4
Population: All treated participants with baseline and post baseline measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491 | Part B - MYH7 - MYK-491 | Part B - TTN - MYK-491 | Part B - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 12 | 11 | 5 | 10 | 8 | 7 | 3
cm/s
  End of treatment period 1: number analyzed (Participants) | 12 | 11 | 4 | 7 | 0 | 0 | 0
  End of treatment period 1 | 0.75 (1.66) | 0.26 (1.62) | -0.05 (1.35) | -0.73 (1.30) |  |  |
  End of treatment period 2: number analyzed (Participants) | 11 | 11 | 5 | 10 | 0 | 0 | 0
  End of treatment period 2 | -0.04 (0.86) | 0.28 (1.59) | 0.84 (1.12) | -0.32 (1.32) |  |  |
  week 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 7 | 3
  week 2 |  |  |  |  | 0.51 (1.43) | -0.84 (1.52) | -0.17 (1.12)
  week 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 6 | 2
  week 6 |  |  |  |  | 0.58 (1.12) | -0.73 (1.94) | -0.10 (2.97)
  week 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 5 | 1
  week 12 |  |  |  |  | 0.60 (1.16) | -0.86 (1.23) | 1.90 (NA) — Insufficient number of participants to calculate standard deviation
  week 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 4 | 0
  week 24 |  |  |  |  | -0.65 (0.76) | -0.75 (0.91) |
  week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  week 36 |  |  |  |  |  | -5.10 (NA) — Insufficient number of participants to calculate standard deviation |
  week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 4 | 0
  week 48 |  |  |  |  | 1.75 (1.32) | -1.50 (1.93) |
  Early termination: number analyzed (Participants) | 1 | 0 | 0 | 0 | 8 | 7 | 3
  Early termination | 0.60 (NA) — Insufficient number of participants to calculate standard deviation |  |  |  | 1.04 (1.65) | 0.04 (1.25) | 1.03 (2.58)

21. Secondary Outcome: Transthoracic Echo (TTE) E/E Prime Average Ratio Change From Baseline
Description: as for outcome 4
Time Frame: as for outcome 4
Population: All treated participants with baseline and post baseline measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: E/E prime ratio
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491 | Part B - MYH7 - MYK-491 | Part B - TTN - MYK-491 | Part B - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 12 | 13 | 5 | 10 | 7 | 7 | 3
E/E prime ratio
  End of treatment period 1: number analyzed (Participants) | 12 | 13 | 4 | 8 | 0 | 0 | 0
  End of treatment period 1 | -2.45 (3.16) | 0.07 (3.67) | -0.20 (4.46) | 0.41 (3.23) |  |  |
  End of treatment period 2: number analyzed (Participants) | 11 | 12 | 5 | 10 | 0 | 0 | 0
  End of treatment period 2 | -2.15 (2.88) | 0.45 (2.99) | -2.16 (3.92) | 1.03 (2.60) |  |  |
  week 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 6 | 3
  week 2 |  |  |  |  | -1.43 (4.37) | -0.03 (4.40) | -0.03 (0.47)
  week 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 6 | 2
  week 6 |  |  |  |  | -1.19 (4.09) | -0.15 (5.41) | 1.25 (1.20)
  week 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 6 | 1
  week 12 |  |  |  |  | -2.24 (1.56) | -0.47 (3.85) | 0.60 (NA) — Insufficient number of participants to calculate standard deviation
  week 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 5 | 0
  week 24 |  |  |  |  | 0.07 (4.67) | -0.66 (4.24) |
  week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  week 36 |  |  |  |  |  | 10.70 (NA) — Insufficient number of participants to calculate standard deviation |
  week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 4 | 0
  week 48 |  |  |  |  | -4.88 (2.38) | -1.00 (3.89) |
  Early termination: number analyzed (Participants) | 1 | 0 | 0 | 0 | 7 | 7 | 3
  Early termination | -0.90 (NA) — Insufficient number of participants to calculate standard deviation |  |  |  | -1.07 (3.30) | -0.51 (3.91) | -0.03 (0.93)

22. Secondary Outcome: Transthoracic Echo (TTE) E/E Prime Lateral Ratio Change From Baseline
Description: as for outcome 4
Time Frame: as for outcome 4
Population: All treated participants with baseline and post baseline measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: E/E prime ratio
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491 | Part B - MYH7 - MYK-491 | Part B - TTN - MYK-491 | Part B - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 11 | 12 | 5 | 10 | 7 | 6 | 3
E/E prime ratio
  End of treatment period 1: number analyzed (Participants) | 11 | 12 | 4 | 8 | 0 | 0 | 0
  End of treatment period 1 | -1.29 (1.72) | -0.08 (3.68) | -1.80 (5.60) | -0.49 (3.94) |  |  |
  End of treatment period 2: number analyzed (Participants) | 11 | 11 | 5 | 10 | 0 | 0 | 0
  End of treatment period 2 | -1.14 (2.23) | 0.12 (2.94) | -3.58 (4.88) | 0.73 (3.93) |  |  |
  week 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 5 | 3
  week 2 |  |  |  |  | -1.07 (2.88) | -1.00 (1.98) | 0.77 (1.42)
  week 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 5 | 2
  week 6 |  |  |  |  | -0.75 (4.23) | -1.34 (2.15) | 1.80 (2.55)
  week 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 5 | 1
  week 12 |  |  |  |  | -2.17 (2.45) | 2.48 (5.43) | 4.00 (NA) — Insufficient number of participants to calculate standard deviation
  week 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 4 | 0
  week 24 |  |  |  |  | -0.45 (3.99) | -0.47 (2.94) |
  week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  week 36 |  |  |  |  |  | 5.00 (NA) — Insufficient number of participants to calculate standard deviation |
  week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 3 | 0
  week 48 |  |  |  |  | -4.08 (3.06) | -1.47 (1.44) |
  Early termination: number analyzed (Participants) | 1 | 0 | 0 | 0 | 7 | 6 | 3
  Early termination | 0.20 (NA) — Insufficient number of participants to calculate standard deviation |  |  |  | -0.91 (3.39) | 0.75 (5.92) | 0.10 (0.62)

23. Secondary Outcome: Transthoracic Echo (TTE) E/E Prime Septal Ratio Change From Baseline
Description: as for outcome 4
Time Frame: as for outcome 4
Population: All treated participants with baseline and post baseline measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: E/E prime ratio
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491 | Part B - MYH7 - MYK-491 | Part B - TTN - MYK-491 | Part B - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 12 | 11 | 5 | 10 | 7 | 7 | 3
E/E prime ratio
  End of treatment period 1: number analyzed (Participants) | 12 | 11 | 4 | 7 | 0 | 0 | 0
  End of treatment period 1 | -3.12 (4.51) | -0.91 (3.78) | 0.65 (2.89) | 1.86 (2.30) |  |  |
  End of treatment period 2: number analyzed (Participants) | 11 | 11 | 5 | 10 | 0 | 0 | 0
  End of treatment period 2 | -1.45 (2.14) | 0.07 (4.00) | -1.38 (2.82) | 1.32 (3.07) |  |  |
  week 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 6 | 3
  week 2 |  |  |  |  | -1.77 (6.75) | 1.50 (9.41) | -0.83 (1.57)
  week 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 6 | 2
  week 6 |  |  |  |  | -1.27 (4.43) | 1.33 (10.61) | 0.65 (0.07)
  week 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 5 | 1
  week 12 |  |  |  |  | -2.27 (3.53) | -1.30 (3.68) | -2.70 (NA) — Insufficient number of participants to calculate standard deviation
  week 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 4 | 0
  week 24 |  |  |  |  | 0.70 (5.41) | -2.03 (7.68) |
  week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  week 36 |  |  |  |  |  | 16.50 (NA) — Insufficient number of participants to calculate standard deviation |
  week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 4 | 0
  week 48 |  |  |  |  | -5.68 (4.89) | 0.05 (7.37) |
  Early termination: number analyzed (Participants) | 1 | 0 | 0 | 0 | 7 | 7 | 3
  Early termination | -2.00 (NA) — Insufficient number of participants to calculate standard deviation |  |  |  | -1.19 (3.67) | -1.19 (4.95) | -0.27 (2.20)

24. Secondary Outcome: Transthoracic Echo (TTE) Ratio of Peak Inflow Velocities in Early and Late Diastole - E/A Change From Baseline
Description: as for outcome 4
Time Frame: as for outcome 4
Population: All treated participants with baseline and post baseline measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: E/A ratio
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491 | Part B - MYH7 - MYK-491 | Part B - TTN - MYK-491 | Part B - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 11 | 11 | 5 | 10 | 6 | 6 | 4
E/A ratio
  End of treatment period 1: number analyzed (Participants) | 11 | 11 | 3 | 10 | 0 | 0 | 0
  End of treatment period 1 | 0.02 (0.16) | -0.01 (0.32) | -0.10 (0.10) | 0.04 (0.11) |  |  |
  End of treatment period 2: number analyzed (Participants) | 11 | 11 | 5 | 10 | 0 | 0 | 0
  End of treatment period 2 | -0.16 (0.40) | -0.08 (0.37) | -0.26 (0.54) | -0.04 (0.15) |  |  |
  week 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 5 | 4
  week 2 |  |  |  |  | 0.07 (0.92) | -0.32 (0.40) | -0.12 (0.21)
  week 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 5 | 2
  week 6 |  |  |  |  | -0.25 (0.45) | -0.58 (0.77) | 0.15 (0.21)
  week 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 5 | 1
  week 12 |  |  |  |  | -0.23 (0.50) | -0.76 (0.70) | 0.20 (NA) — Insufficient number of participants to calculate standard deviation
  week 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 4 | 0
  week 24 |  |  |  |  | 0.00 (0.10) | -0.53 (0.78) |
  week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  week 36 |  |  |  |  |  | 0.20 (NA) — Insufficient number of participants to calculate standard deviation |
  week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 3 | 0
  week 48 |  |  |  |  | -0.40 (0.52) | -0.77 (0.85) |
  Early termination: number analyzed (Participants) | 1 | 0 | 0 | 0 | 5 | 6 | 3
  Early termination | 0.70 (NA) — Insufficient number of participants to calculate standard deviation |  |  |  | -0.10 (0.32) | -0.37 (0.52) | 0.17 (0.06)

25. Secondary Outcome: Transthoracic Echo (TTE) Left Atrial Minimum Volume (LAminV) Change From Baseline
Description: as for outcome 4
Time Frame: as for outcome 4
Population: All treated participants with baseline and post baseline measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491 | Part B - MYH7 - MYK-491 | Part B - TTN - MYK-491 | Part B - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 12 | 14 | 4 | 9 | 8 | 7 | 3
mL
  End of treatment period 1: number analyzed (Participants) | 12 | 14 | 4 | 9 | 0 | 0 | 0
  End of treatment period 1 | -2.545 (4.182) | -0.374 (8.947) | -3.663 (9.552) | -0.563 (3.670) |  |  |
  End of treatment period 2: number analyzed (Participants) | 11 | 14 | 4 | 9 | 0 | 0 | 0
  End of treatment period 2 | -3.985 (5.681) | 0.049 (8.529) | -3.993 (5.672) | -2.866 (6.613) |  |  |
  week 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 7 | 3
  week 2 |  |  |  |  | 0.509 (11.279) | -3.807 (9.917) | 2.817 (8.224)
  week 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 6 | 2
  week 6 |  |  |  |  | 3.430 (9.313) | -10.938 (22.821) | 1.680 (5.374)
  week 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 6 | 1
  week 12 |  |  |  |  | -3.409 (13.577) | -13.953 (24.798) | 9.950 (NA) — Insufficient number of participants to calculate standard deviation
  week 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 5 | 0
  week 24 |  |  |  |  | -2.858 (16.826) | -5.214 (32.177) |
  week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  week 36 |  |  |  |  |  | -16.410 (NA) — Insufficient number of participants to calculate standard deviation |
  Week 42: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Week 42 |  |  |  |  |  | -27.640 (NA) — Insufficient number of participants to calculate standard deviation |
  week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 4 | 0
  week 48 |  |  |  |  | -7.560 (7.287) | -19.843 (24.404) |
  Early termination: number analyzed (Participants) | 1 | 0 | 0 | 0 | 8 | 7 | 3
  Early termination | 12.030 (NA) — Insufficient number of participants to calculate standard deviation |  |  |  | 1.313 (13.248) | -4.793 (19.027) | 10.607 (3.279)

26. Secondary Outcome: Transthoracic Echo (TTE) Left Atrial Maximum Volume Index (LAmaxVi) Change From Baseline
Description: as for outcome 4
Time Frame: as for outcome 4
Population: All treated participants with baseline and post baseline measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491 | Part B - MYH7 - MYK-491 | Part B - TTN - MYK-491 | Part B - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 12 | 14 | 4 | 9 | 8 | 7 | 3
mL/m^2
  End of treatment period 1: number analyzed (Participants) | 12 | 14 | 4 | 9 | 0 | 0 | 0
  End of treatment period 1 | -0.6427 (5.0007) | 0.9860 (7.1462) | -0.6320 (9.1208) | -0.0084 (2.4459) |  |  |
  End of treatment period 2: number analyzed (Participants) | 11 | 14 | 4 | 9 | 0 | 0 | 0
  End of treatment period 2 | -0.3419 (4.2365) | 1.1617 (6.0815) | -1.1870 (7.2047) | -0.2139 (2.5533) |  |  |
  week 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 7 | 3
  week 2 |  |  |  |  | 0.1346 (6.4456) | -0.1818 (5.1802) | 2.3315 (9.2253)
  week 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 6 | 2
  week 6 |  |  |  |  | 1.1887 (4.2647) | -5.5545 (13.4164) | -0.5969 (10.1570)
  week 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 6 | 1
  week 12 |  |  |  |  | -1.9834 (9.0618) | -7.1717 (14.8684) | 7.8293 (NA) — Insufficient number of participants to calculate standard deviation
  week 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 5 | 0
  week 24 |  |  |  |  | -2.3145 (11.3192) | -1.8423 (17.8500) |
  week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 2 | 0
  week 36 |  |  |  |  |  | -13.3385 (3.1173) |
  Week 42: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Week 42 |  |  |  |  |  | -11.7208 (NA) — Insufficient number of participants to calculate standard deviation |
  week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 4 | 0
  week 48 |  |  |  |  | -2.4524 (3.4679) | -11.2887 (15.6892) |
  Early termination: number analyzed (Participants) | 1 | 0 | 0 | 0 | 8 | 7 | 3
  Early termination | 8.1892 (NA) — Insufficient number of participants to calculate standard deviation |  |  |  | -0.0097 (6.8537) | -1.4975 (9.7454) | 6.5957 (3.9106)

27. Secondary Outcome: Transthoracic Echo (TTE) Left Atrial Emptying Fraction (LAEF) Change From Baseline
Description: as for outcome 4
Time Frame: as for outcome 4
Population: All treated participants with baseline and post baseline measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491 | Part B - MYH7 - MYK-491 | Part B - TTN - MYK-491 | Part B - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 12 | 14 | 4 | 9 | 8 | 7 | 3
Percent change
  End of treatment period 1: number analyzed (Participants) | 12 | 14 | 4 | 9 | 0 | 0 | 0
  End of treatment period 1 | 5.617 (13.459) | 4.675 (12.173) | 2.687 (26.913) | 2.489 (10.953) |  |  |
  End of treatment period 2: number analyzed (Participants) | 11 | 14 | 4 | 9 | 0 | 0 | 0
  End of treatment period 2 | 15.504 (18.234) | 9.870 (15.019) | 8.102 (21.513) | 9.655 (14.789) |  |  |
  week 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 7 | 3
  week 2 |  |  |  |  | -1.903 (19.042) | 15.609 (10.759) | 1.058 (6.753)
  week 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 6 | 2
  week 6 |  |  |  |  | -9.410 (20.950) | 21.196 (24.108) | -7.265 (24.267)
  week 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 6 | 1
  week 12 |  |  |  |  | 5.089 (17.898) | 24.306 (30.693) | -6.694 (NA) — Insufficient number of participants to calculate standard deviation
  week 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 5 | 0
  week 24 |  |  |  |  | 6.522 (23.635) | 19.181 (31.252) |
  week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  week 36 |  |  |  |  |  | 2.595 (NA) — Insufficient number of participants to calculate standard deviation |
  Week 42: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Week 42 |  |  |  |  |  | 43.996 (NA) — Insufficient number of participants to calculate standard deviation |
  week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 4 | 0
  week 48 |  |  |  |  | 23.815 (26.494) | 27.568 (24.279) |
  Early termination: number analyzed (Participants) | 1 | 0 | 0 | 0 | 8 | 7 | 3
  Early termination | -7.060 (NA) — Insufficient number of participants to calculate standard deviation |  |  |  | -0.711 (30.276) | 11.267 (25.412) | -6.924 (11.148)

28. Secondary Outcome: Transthoracic Echo (TTE) Left Atrial Function Index (LAFI) Change From Baseline
Description: Baseline is defined as the last non-missing result prior to the first dose of study medication. for part B, baseline is defined as visit 1B regardless of rescreening. Treatment periods 1 and 2 are 5 to 8 days. Higher LAFI values are considered better left atrial function while lower LFAI values may indicate left atrial dysfunction.
Time Frame: as for outcome 4
Population: All treated participants with baseline and post baseline measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Part A - MYH7 - MYK-491 | Part A - TTN - MYK-491 | Part A - DCM-Genetic - MYK-491 | Part A - DCM-Non Genetic - MYK-491 | Part B - MYH7 - MYK-491 | Part B - TTN - MYK-491 | Part B - DCM-Non Genetic - MYK-491
Number analyzed (Participants) | 12 | 14 | 4 | 9 | 8 | 7 | 3
Index
  End of treatment period 1: number analyzed (Participants) | 12 | 14 | 4 | 9 | 0 | 0 | 0
  End of treatment period 1 | 5.2299 (5.3847) | 1.6645 (11.9891) | -0.4600 (1.6721) | 0.3524 (5.0864) |  |  |
  End of treatment period 2: number analyzed (Participants) | 11 | 14 | 4 | 9 | 0 | 0 | 0
  End of treatment period 2 | 11.1434 (10.5287) | 6.8482 (13.2805) | 1.6243 (5.5803) | 3.6366 (6.4861) |  |  |
  week 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 7 | 3
  week 2 |  |  |  |  | 4.1989 (10.0937) | 5.6654 (7.6211) | -10.2619 (21.2810)
  week 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 6 | 2
  week 6 |  |  |  |  | 0.7215 (23.0068) | 9.9039 (8.9999) | 1.3624 (15.4676)
  week 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 6 | 1
  week 12 |  |  |  |  | 5.3578 (14.5382) | 8.4149 (7.3469) | -22.1266 (NA) — Insufficient number of participants to calculate standard deviation
  week 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 5 | 0
  week 24 |  |  |  |  | -4.8648 (19.3724) | 8.1890 (8.8584) |
  week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 2 | 0
  week 36 |  |  |  |  |  | 8.6083 (8.6083) |
  week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 4 | 0
  week 48 |  |  |  |  | 6.3041 (18.4543) | 12.8222 (14.0703) |
  Early termination: number analyzed (Participants) | 1 | 0 | 0 | 0 | 8 | 7 | 3
  Early termination | -11.0849 (NA) — Insufficient number of participants to calculate standard deviation |  |  |  | 0.3925 (23.9350) | 2.4252 (10.4948) | -20.4736 (4.7293)

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious adverse events, and other adverse events are from first dose until the end of the study visit for the participant (Up to approximately 115 weeks)
Description: The participant will receive 25mg BID dose in Part A Treatment Period 1 and then the same participant will be up-titrated to 50mg BID or down-titrated to 10mg BID in Part A Treatment Period 2. The Part B starting dose can be either 5 mg BID, 10 mg BID, 25 mg BID, 50 mg BID, or 75 mg BID, and then the same participant will be up-titrated or down-titrated to a dose based on systolic ejection time.
Groups:
- Part A - MYH7 - MYK-491 25 mg BID; Part B - MYH7 - MYK-491 25 mg BID: Participants with MYH7 variant received 25 mg BID Danicamtiv
- Part A - TTN - MYK-491 25 mg BID: Participants with TTN variant received 25 mg BID Danicamtiv
- Part A - DCM-Genetic - MYK-491 25 mg BID: Participants with DCM-Genetic variant received 25 mg BID Danicamtiv
- Part A - DCM-Non Genetic - MYK-491 25 mg BID: Participants with DCM-Non genetic variant received 25 mg BID Danicamtiv
- Part A - MYH7 - MYK-491 50 mg BID; Part B - MYH7 - MYK-491 50 mg BID: Participants with MYH7 variant received 50 mg BID Danicamtiv
- Part A - TTN - MYK-491 50 mg BID; Part B - TTN - MYK-491 50 mg BID: Participants with TTN variant received 50 mg BID Danicamtiv
- Part A - DCM-Genetic - MYK-491 50 mg BID: Participants with DCM-Genetic variant received 50 mg BID Danicamtiv
- Part A - DCM-Non Genetic - MYK-491 50 mg BID; Part B - DCM-Non Genetic - MYK-491 50 mg BID: Participants with DCM-Non genetic variant received 50 mg BID Danicamtiv
- Part A - DCM-Genetic - MYK-491 10 mg BID: Participants with DCM-Genetic variant received 10 mg BID Danicamtiv
- Part A - DCM-Non Genetic - MYK-491 10 mg BID: Participants with DCM-Non genetic variant received 10 mg BID Danicamtiv
- Part B - MYH7 - MYK-491 75 mg BID: Participants with MYH7 variant received 75 mg BID Danicamtiv
- Part B - TTN - MYK-491 75 mg BID: Participants with TTN variant received 75 mg BID Danicamtiv
- Part B - DCM-Non Genetic - MYK-491 75 mg BID: Participants with DCM-Non genetic variant received 75 mg BID Danicamtiv
Arm/Group | Part A - MYH7 - MYK-491 25 mg BID | Part A - TTN - MYK-491 25 mg BID | Part A - DCM-Genetic - MYK-491 25 mg BID | Part A - DCM-Non Genetic - MYK-491 25 mg BID | Part A - MYH7 - MYK-491 50 mg BID | Part A - TTN - MYK-491 50 mg BID | Part A - DCM-Genetic - MYK-491 50 mg BID | Part A - DCM-Non Genetic - MYK-491 50 mg BID | Part A - DCM-Genetic - MYK-491 10 mg BID | Part A - DCM-Non Genetic - MYK-491 10 mg BID | Part B - MYH7 - MYK-491 25 mg BID | Part B - MYH7 - MYK-491 50 mg BID | Part B - TTN - MYK-491 50 mg BID | Part B - DCM-Non Genetic - MYK-491 50 mg BID | Part B - MYH7 - MYK-491 75 mg BID | Part B - TTN - MYK-491 75 mg BID | Part B - DCM-Non Genetic - MYK-491 75 mg BID
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/14 | 0/5 | 0/10 | 0/12 | 0/14 | 0/4 | 0/9 | 0/1 | 0/1 | 0/1 | 0/4 | 0/4 | 0/1 | 0/5 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14 | 0/5 | 0/10 | 0/12 | 0/14 | 0/4 | 0/9 | 0/1 | 0/1 | 0/1 | 1/4 | 1/4 | 0/1 | 0/5 | 2/4 | 1/3
Other Adverse Events (participants affected / at risk) | 5/12 | 3/14 | 1/5 | 2/10 | 5/12 | 5/14 | 2/4 | 2/9 | 0/1 | 0/1 | 1/1 | 3/4 | 3/4 | 0/1 | 5/5 | 4/4 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A - MYH7 - MYK-491 25 mg BID (N=12) | Part A - TTN - MYK-491 25 mg BID (N=14) | Part A - DCM-Genetic - MYK-491 25 mg BID (N=5) | Part A - DCM-Non Genetic - MYK-491 25 mg BID (N=10) | Part A - MYH7 - MYK-491 50 mg BID (N=12) | Part A - TTN - MYK-491 50 mg BID (N=14) | Part A - DCM-Genetic - MYK-491 50 mg BID (N=4) | Part A - DCM-Non Genetic - MYK-491 50 mg BID (N=9) | Part A - DCM-Genetic - MYK-491 10 mg BID (N=1) | Part A - DCM-Non Genetic - MYK-491 10 mg BID (N=1) | Part B - MYH7 - MYK-491 25 mg BID (N=1) | Part B - MYH7 - MYK-491 50 mg BID (N=4) | Part B - TTN - MYK-491 50 mg BID (N=4) | Part B - DCM-Non Genetic - MYK-491 50 mg BID (N=1) | Part B - MYH7 - MYK-491 75 mg BID (N=5) | Part B - TTN - MYK-491 75 mg BID (N=4) | Part B - DCM-Non Genetic - MYK-491 75 mg BID (N=3)
Arrhythmic storm (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A - MYH7 - MYK-491 25 mg BID (N=12) | Part A - TTN - MYK-491 25 mg BID (N=14) | Part A - DCM-Genetic - MYK-491 25 mg BID (N=5) | Part A - DCM-Non Genetic - MYK-491 25 mg BID (N=10) | Part A - MYH7 - MYK-491 50 mg BID (N=12) | Part A - TTN - MYK-491 50 mg BID (N=14) | Part A - DCM-Genetic - MYK-491 50 mg BID (N=4) | Part A - DCM-Non Genetic - MYK-491 50 mg BID (N=9) | Part A - DCM-Genetic - MYK-491 10 mg BID (N=1) | Part A - DCM-Non Genetic - MYK-491 10 mg BID (N=1) | Part B - MYH7 - MYK-491 25 mg BID (N=1) | Part B - MYH7 - MYK-491 50 mg BID (N=4) | Part B - TTN - MYK-491 50 mg BID (N=4) | Part B - DCM-Non Genetic - MYK-491 50 mg BID (N=1) | Part B - MYH7 - MYK-491 75 mg BID (N=5) | Part B - TTN - MYK-491 75 mg BID (N=4) | Part B - DCM-Non Genetic - MYK-491 75 mg BID (N=3)
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chalazion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site rash (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device inappropriate shock delivery (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Initial insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/93/NCT04572893/Prot_SAP_000.pdf